CLINICAL TRIAL: NCT06225700
Title: Clinical Validation of Novel Malaria Diagnostic Tools for Point-of-Care Testing
Brief Title: Clinical Validation of Novel Malaria Diagnostic Tools for POC Point-of-Care Testing
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Australian Government (Unknown)
Responsible Party: Sponsor
Other Study IDs: MA017
Record Dates: First submitted 2023-01-23; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-03

CONDITIONS: Malaria; Diagnoses Disease; RDT
Keywords: Malaria, diagnostics
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Capillary blood, Venous blood, Foot odour
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to perform a performance evaluation of novel diagnostic tools for detecting malaria in malaria-endemic countries. At the beginning of 2022, FIND launched a call for innovation with the distinct aim to identify malaria innovations that have the potential to address the technical and operational limitations of current malaria RDTs, particularly in view of the emergence of P. falciparum parasites with hrp2/3 deletions, the need for improved tools to identify all Plasmodium species and/or the need for improved surveillance.

This study will generate valuable data on the performance of these novel non-HRP2-based tests and inform FIND and developers on technical and operational assay optimization requirements for accelerated access of these tools to market.

DETAILED DESCRIPTION:
This study aims to support product development efforts towards novel malaria diagnostics not HRP2-based by providing early-stage technology developers with valuable information on performance and basic feasibility data that can help to accelerate development. The WHO now recommends that where pfhrp2/3 gene deletions are reported (within countries or in neighboring countries), representative baseline surveys are to be conducted among suspected cases. If >5% of false negative RDT results are attributed to these deletions, a change in RDT is necessary. Plasmodium lactate dehydrogenase (pLDH), appears as a good alternative to HRP2 as it is an essential protein expressed by all human-infecting Plasmodium species. However, pLDH-based RDTs have shown to perform poorly at low parasitaemia, which is common among patients infected with P. vivax, P. malariae and P. ovale species as well as in asymptomatic infections. Thus, RDTs not based on HRP2 are limited; moreover, WHO prequalified ones that can detect and distinguish between Plasmodium falciparum and Plasmodium vivax are non-existent. The current malaria diagnostic landscape demands more innovation supporting and accelerating the development of new malaria diagnostic tools that that tackle these emerging issues.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years or older
* Presenting at the study site with symptoms and signs suggestive of malaria
* Freely agreeing to participate by signing an informed consent form (adults aged 18 and older and parent/legal guardian of a child) and providing assent (children aged 13-17)
* Willing to provide venous blood sample and other samples such as foot odour.

Exclusion Criteria:

* Presence of symptoms and signs of severe disease and/or central nervous system infections, as defined by WHO guidelines

Participants are excluded from the foot odour collection if the following exclusion criteria apply:

* Skin lesions on the feet
* Infected skin on the feet
* Infected toenails

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in multiple primary health care facilities (e.g., health posts, health centres) where malaria diagnosis is provided on a routine basis in malaria-endemic Rwanda. The study population will be patients with symptoms suggestive of malaria seeking clinical care in a health facility.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Performance of nPOC | 3 months
  Point estimates of clinical performance characteristics (sensitivity, specificity, NPV, PPV, and DOR) with 95% confidence intervals of nPOC using nPCR as reference for detecting malaria in patients with symptoms suggestive of malaria.

SECONDARY OUTCOMES:
Performance of LM | 3 months
  Point estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV, and DOR) of light microscopy using nPCR as reference for detecting malaria in patients with symptoms suggestive of malaria
Performance of comparator RDT | 3 months
  Point estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV, and DOR) of the comparator tests using nPCR as reference for detecting malaria in patients with symptoms suggestive of malaria
Comparison between nPOC [Truenat® Malaria Pv/Pf; Truenat® Malaria Pv/Pf Hi-Sens; Humasis Hs-Malaria P.f/Pan test, Hemozoin Imager] and LM | 3 months
  Comparison between the clinical performance of nPOC and light microscopy
Comparison between Hemozoin Imager and comparator RDT | 3 months
  Comparison between the clinical performance of between the clinical performance of Hemozoin Imager and comparator rapid diagnostic test [SD Bioline Combo/ First Response].
  The percentage difference between the clinical performance characteristics of nPOC and comparator RDT with 95% confidence intervals using Tango's score method.
Comparison of Truenat Pv/Pf and Truenat Pv/Pf High-Sens | 3 months
  Comparison between clinical performance of Truenat® Pv/Pf and Truenat® Pv/Pf Hi-Sens.
  The percentage difference between the clinical performance characteristics of Truenat® Pv/Pf and Truenat® Pv/Pf Hi-Sens with 95% confidence intervals using Tango's score method.
Comparison between Truenat Pv/Pf and Truenat Pv/Pf High-Sens and Realstar | 3 months
  Comparison between the clinical performance of Truenat® Pv/Pf and Truenat® Pv/Pf Hi-Sens with that of RealStar® Malaria Screen & Type PCR Kit 1.0.
  The percentage difference between the clinical performance characteristics of the Truenat® tests (Truenat® Pv/Pf and Truenat® Pv/Pf Hi-Sens) and RealStar® Malaria Screen & Type PCR Kit 1.0 with 95% confidence intervals using Tango's score method.
Foot odour collection | 3 months
  The number of volatile organic compound (foot odour samples) from Plasmodium positive and negative febrile patients that have been collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Stansile, Kigali, Rwanda

REFERENCES:
- [Background] World Health Organization. "False-Negative RDT Results and P. Falciparum Histidine-Rich Protein 2/3 Gene Deletions." Global Malaria Programme, July 2019.
- [Background] World Health Organization, 2018. Malaria Rapid Diagnostic Test Performance; Summary results of WHO product testing of malaria RDTs: round 1-8 (2008-2018). Geneva.
- [Background] World Health Organization, 2015. Control and Elimination of Plasmodium Vivax Malaria: A Technical Brief. Geneva: WHO Press.